CLINICAL TRIAL: NCT07079969
Title: Effects of Photobiomodulation and Topical Diclofenac on Inflammation and Pain in Knee Osteoarthritis
Brief Title: Effects of Photobiomodulation and Topical Diclofenac on Inflammation and Pain in Knee Osteoarthritis (EPIC-KO)
Acronym: EPIC-KO
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IRB202501000
Record Dates: First submitted 2025-07-09; First posted 2025-07-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-07

CONDITIONS: Knee Pain Chronic
MeSH Terms: interventions — Low-Level Light Therapy; Phototherapy; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- PBM Only (Experimental): Participants will receive placebo topical cream (identical in appearance to diclofenac sodium 1% gel), applied at a dose of 4 grams to the affected knee during each treatment session. They will also receive active photobiomodulation therapy (PBM) using an FDA-cleared near-infrared device. PBM will be administered approximately 10 minutes after placebo cream application. Both treatments will be delivered in six sessions over a 2-3 week period, at a frequency of 2-3 times per week.
  Interventions: Device: Photobiomodulation therapy (PBM) device; Drug: Placebo topical cream
- Diclofenac only (Experimental): Participants will receive diclofenac sodium 1% topical cream, applied at a dose of 4 grams to the affected knee during each treatment session. They will also receive sham PBM using a device identical in appearance to the active PBM device but without therapeutic light output. Sham PBM will be administered approximately 10 minutes after diclofenac cream application. Both treatments will be delivered in six sessions over 2-3 weeks, at a frequency of 2-3 times per week.
  Interventions: Device: Sham PBM device; Drug: Diclofenac Sodium 1 % Topical Cream
- Combined (Experimental): Participants will receive diclofenac sodium 1% topical cream, applied at a dose of 4 grams to the affected knee during each treatment session. They will also receive active PBM using the same device and parameters described above. PBM will be administered approximately 10 minutes after diclofenac cream application. Both treatments will be delivered in six sessions over 2-3 weeks, at a frequency of 2-3 times per week.
  Interventions: Device: Photobiomodulation therapy (PBM) device; Drug: Diclofenac Sodium 1 % Topical Cream
- Double placebo (Placebo Comparator): Participants will receive placebo topical cream, applied at a dose of 4 grams to the affected knee during each treatment session. They will also receive sham PBM using a visually identical device that does not emit therapeutic light. Sham PBM will be administered approximately 10 minutes after placebo cream application. Both treatments will be delivered in six sessions over 2-3 weeks, at a frequency of 2-3 times per week.
  Interventions: Device: Sham PBM device; Drug: Placebo topical cream

INTERVENTIONS:
Device: Photobiomodulation therapy (PBM) device — FDA-cleared near-infrared PBM device delivering therapeutic light to the affected knee. Administered once per session, approximately 10 minutes after topical application, in six sessions over 2-3 weeks (2-3 times per week).
  Other Names: light therapy
  Arms: Combined; PBM Only
Device: Sham PBM device — Identical in appearance to the active PBM device but emits no therapeutic light. Administered once per session, approximately 10 minutes after topical application, in six sessions over 2-3 weeks.
  Other Names: placebo light therapy
  Arms: Diclofenac only; Double placebo
Drug: Diclofenac Sodium 1 % Topical Cream — Topical nonsteroidal anti-inflammatory drug applied at a dose of 4 grams to the affected knee, once per session, immediately before PBM/sham PBM. Used in six sessions over 2-3 weeks.
  Other Names: Voltaren; NSAID topical cream
  Arms: Combined; Diclofenac only
Drug: Placebo topical cream — Inert cream matching the appearance of diclofenac sodium 1% gel. Applied at 4 grams to the affected knee, once per session, immediately before PBM/sham PBM. Used in six sessions over 2-3 weeks
  Other Names: Vehicle cream
  Arms: Double placebo; PBM Only

SUMMARY:
This study aims to compare the effects of combined treatments-dual-wavelength photobiomodulation (PBM) with or without topical diclofenac-on inflammation, pain, and joint function in patients with knee osteoarthritis (OA). It also seeks to determine the synergistic effect of PBM plus topical diclofenac on inflammatory markers, pain scores, and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed knee osteoarthritis (OA) based on the American College of Rheumatology (ACR) criteria with symptomatic pain for ≥ 3 months
* Average knee-pain intensity ≥ 30/100 on both the Daily Symptom Diary (DSD) run-in and CATI
* Age ≥ 50 years
* Ability to give informed consent, attend visits, and complete ≥ 4 of 7 DSD entries pre-randomization
* Capacity to perform all study tasks (Timed Up-and-Go, knee OA assessments, blood draw, questionnaires, etc)

Exclusion Criteria:

Systemic and Rheumatic Disease

* Active systemic rheumatic condition (e.g., rheumatoid arthritis, systemic lupus erythematosus)
* Fibromyalgia with pain outside the knee that is equal to or worse than knee pain

Musculoskeletal History

* Clinically significant surgery on the index knee (e.g., arthroplasty, osteotomy)
* Knee surgery within the past 6 weeks
* Intra-articular injection to the index knee within the past 14 days

Medication Use

* Daily opioid therapy
* Hypersensitivity or allergy to diclofenac, other NSAIDs, or PBM
* Use of centrally acting sodium-channel blockers or NMDA-receptor antagonists
* New prescription or OTC analgesic, non-pharmacologic pain therapy, investigational drug, chemotherapy, or radiation therapy initiated ≤ 30 days before screening
* Clinically significant drug interaction between topical diclofenac and concomitant medications per Drugs.com Drug Interaction Checker

Cardiovascular Safety

* Uncontrolled hypertension (SBP > 150 mmHg or DBP > 95 mmHg)
* Unstable or activity-limiting cardiovascular or peripheral arterial disease

Neurological and Psychiatric Conditions

* Diagnosed neurological disorder (e.g., Parkinson's disease, multiple sclerosis, epilepsy)
* History or evidence of stroke or moderate-severe traumatic brain injury
* Serious psychiatric illness requiring hospitalization within the past 12 months
* Active suicidal ideation
* Current substance-use disorder or past hospitalization for substance-use treatment

Dermatologic Conditions

* Compromised skin integrity at or near the treatment site (e.g., open wounds, active rash, dermatitis, burns, ulcers, eczema, infection) interfering with topical treatment or PBM

Renal Function

* Severe renal impairment
* History of acute kidney injury within the past 6 months

Hepatic Function

* Active liver disease or elevated liver enzymes
* Known moderate to severe hepatic impairment
* Acute or chronic liver disease such as hepatitis

Other Metabolic Conditions

* Uncontrolled diabetes
* Diabetes-related complications (e.g., peripheral neuropathy, severe nephropathy, chronic ulcers at treatment site)
* Active peptic ulcers or history of recurrent peptic ulcers with complications (e.g., bleeding, perforation)
* Current use of anticoagulants with a history of gastrointestinal ulceration

Other Pain Conditions

* Chronic pain at another body site more severe than knee pain

General Health and Cognition

* Severe circulatory disorder
* Pregnancy or lactation
* Cognitive impairment that precludes informed consent or task participation

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Pain Intensity (Numeric Rating Scale) | Baseline (Visit 0) to Final Follow-up (Visit 7; approximately 3-4 weeks after baseline)
  Knee pain will be assessed using the 0-10 Numeric Rating Scale (NRS), where 0 indicates no pain and 10 indicates the worst imaginable pain. Assessments will be conducted at baseline (V0) and at the final follow-up visit, one week after the last treatment session.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
This is a small, internally funded pilot study intended to assess feasibility and preliminary outcomes. IPD sharing is not planned at this stage.